CLINICAL TRIAL: NCT03732885
Title: Crestal Maxillary Sinus Floor Elevation Using Osseodensification Drills (Densah Burs) Versus Summers Osteotomes
Brief Title: Maxillary Sinus Floor Elevation Using DENSAH Burs Versus Summers Osteotomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sohaib Mohamed Alzamzamy Mohamed Elsheikh, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NCT035
Record Dates: First submitted 2018-10-30; First posted 2018-11-07 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Implant Tissue Failure
Keywords: Sinus; Stability; Bone gain; Osseodensification
MeSH Terms: conditions — Fistula

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- densah burs drilling group (Experimental): maxillary sinus floor elevation during implant placement using Densah burs
  Interventions: Device: densah burs osseo densification drills
- Summers osteotomes (Experimental): maxillary sinus floor elevation during implant placement using Summer's Osteotomes
  Interventions: Device: Summer's Osteotomes

INTERVENTIONS:
Device: densah burs osseo densification drills — maxillary sinus floor elevation during implant placement using Densah burs
  Arms: densah burs drilling group
Device: Summer's Osteotomes — maxillary sinus floor elevation during implant placement using Summer's Osteotomes
  Arms: Summers osteotomes

SUMMARY:
To investigate the efficacy of osseodensification drills (Densah bure) as a new closed sinus lift tool and to compare the effect of it in bone gaine versus traditional osteotomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with partially edentulous in the posterior area of the maxilla, with a residual ridge that allowed insertion of ≤8 mm length implants.
* both sexes.
* No intraoral soft and hard tissue pathology
* No systemic condition that contraindicate implant placement.

Exclusion Criteria:

* Sinus pathology.
* Heavy smokers more than 20 cigarettes per day.
* Patients with systemic disease that may affect normal healing.
* Psychiatric problems.
* Disorders to implant are related to history of radiation therapy to the head and neck neoplasia, or bone augmentation to implant site.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2019-04-15 (Estimated); Study Completion 2019-07-15 (Estimated)

PRIMARY OUTCOMES:
implant stability | 6 months after surgery
  measurement of implant stability using the Ostell

SECONDARY OUTCOMES:
bone gain | 6 months after surgery
  measurement of bone gain around implant using cone-beam computed tomography CBCT

CONTACTS AND LOCATIONS:
Locations (1):
- Sohaib M Elsheikh, Cairo, Egypt